CLINICAL TRIAL: NCT03463200
Title: The Influence of Kinesio Taping on Back Muscle Fatigue of Low Back Pain Patients
Brief Title: KT on Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Associate Professor and Researcher, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LBM2018
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
Keywords: bandage; low back pain; muscle fatigue; electromyography
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): It will not apply any tape.
- Experimental group 1 (Experimental): Apply the KT with tension in the erector spine muscles.
  Interventions: Other: Functional elastic tape tensioned
- Experimental group 2 (Experimental): Apply the KT without tension in the erector spine muscles.
  Interventions: Other: Functional elastic tape non-tensioned
- Experimental group 3 (Experimental): Apply Micropore tape in the erector spine muscles.
  Interventions: Other: Rigid Tape

INTERVENTIONS:
Other: Functional elastic tape tensioned — Application of Kinesio Taping with tension in the erector spine muscles.
  Other Names: Kinesio Taping with tension
  Arms: Experimental group 1
Other: Functional elastic tape non-tensioned — Application of Kinesio Taping without tension in the erector spine muscles.
  Other Names: Kinesio Taping without tension
  Arms: Experimental group 2
Other: Rigid Tape — Application of Micropore tape in the erector spine muscles.
  Other Names: Micropore Tape
  Arms: Experimental group 3

SUMMARY:
This study aim evaluates the effect of Kinesio Taping (KT) on back muscle fatigue of low back pain patients, analysing the electromyography activity of longissimus muscle (median frequency) and the sustained time during a fatigue test (Ito test).

DETAILED DESCRIPTION:
Individuals with low back pain usually have poor back muscles endurance, which may be improved with the application of Kinesio Taping. The aim of this study is evaluate the effect of Kinesio Taping on back muscle fatigue of low back pain patients. Sixty-four women, between 18 to 50 years old, with chronic nonspecific Low Back Pain will attend this study. They will be randomly assigned in four different groups: control group (CG), KT with tension group (KTT), KT no tension group (KTNT) and Micropore® group (MP) and submitted to three evaluations: pre, three and ten days after intervention, analysing the electromyography activity of longissimus muscle and the sustained time during a fatigue test. The variables analysed during the evaluations will be median frequency (MP) slope of longuissimus muscle and sustained time during the Ito test.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 50 years of age with chronic nonspecific low back pain for more than three months.

Exclusion Criteria:

* Serious spinal pathologies (fractures, tumors, and inflammatory pathologies such as ankylosing spondylitis);
* Nerve root compromise (disc herniation and spondylolisthesis with neurological compromise, spinal stenosis, and others);
* Fibromyalgia
* Corticosteroid treatment in the previous two weeks;
* Antiinflammatory treatment in the previous 24 hours;
* Contraindications to the use of Kinesio Taping (allergy or intolerance);
* Score of two or less on Visual Analogue Scale of the first day;
* Pregnancy;
* Previous Kinesio Tape therapy on lumbar.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Median frequency | Change from baseline median frequency at three days after the application of the tape.
  Median frequency slope measured my electromyography

SECONDARY OUTCOMES:
Median frequency | Change from baseline median frequency at ten days after the application of the tape.
  Median frequency slope measured my electromyography
Sustained muscle fatigue time | Change from baseline sustained time at three days after the application of the tape.
  Sustained time during a fatigue test
Sustained muscle fatigue time | Change from baseline sustained time at ten days after the application of the tape.
  Sustained time during a fatigue test

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No